CLINICAL TRIAL: NCT02294500
Title: Multicenter Cohort Study to Evaluate and to Protect Ovarian Function and Reproductive Function
Brief Title: Cohort Study to Evaluate Ovarian Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shixuan Wang (Other)
Collaborators: Huazhong University of Science and Technology (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Zhengzhou University (Other); Shanghai Jiao Tong University School of Medicine (Other); Xinjiang Medical University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Shixuan Wang, Study Chairman, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: OA-1-female
Record Dates: First submitted 2014-09-10; First posted 2014-11-19 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve; Menopausal Syndrome; Sexual Function and Fertility Disorders; Cardiovascular Diseases
Keywords: ovarian function; female; Genital Function
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Our biospecimen included blood, serum, plasma and other body fluid and tissues
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will collect the clinical and biological data of the patients, the investigators could further analyse and identify the risk factors and optimize clinical treatment method. Besides, population-based healthy people with informed consent are also collected.

DETAILED DESCRIPTION:
Menopause is the last step in the process of ovarian ageing. Decrease in follicle numbers dictates the onset of cycle irregularity and the cessation of menses. At the same time, decaying in oocyte quality contributes to the gradual decline in fertility. Endocrine changes mainly depend on the decline in the negative feedback by ovarian factors at the hypothalamo-pituitary unit. The declining antral follicle cohort(AFC) with age first results in gradually elevated FSH levels. The gradual decline in the size of AFC is best represented by decreasing levels of anti-Mullerian hormone. The identification of women who have severely decreased ovarian reserve is clinically relevant. Ovarian reserve tests have appeared to be fairly accurate in predicting response to ovarian stimulation in the assisted reproductive technology (ART) setting. The capacity to predict the chances for spontaneous pregnancy or pregnancy after ART appears very limited. As menopause and the preceding decline in oocyte quality seem to have a fixed time interval, tests that predict the age at menopause may be useful to assess individual reproductive lifespan like genetic studies, ovarian ageing mechanism studies and epigenetic studies.

Heart disease remains a major cause of death among women in China. We focuses on physiologic endogenous sex steroid levels and heart disease especially for CAD among postmenopausal women with natural or surgical menopause. Now there are more and more reasons to seek evidence for associations of circulating estrogen or other endogenous sex steroid levels and CAD. In the future, we design a cohort study to confirm whether ovarian sex steroid hormonal changes is associated with CAD postmenopausal women, or there may be other components explaining the gender differences in CAD patterns.

Premature ovarian failure(POF), is a disorder of infertility characterized by amenorrhoea, low estrogen levels and increased gonadotropin levels in women aged <40 years. POF is the result of premature exhaustion of the follicle pool or can be attributed to follicular dysfunction, for example, owing to mutations in the FSH receptor or steroidogenic cell autoimmunity. Moreover, advances in cancer therapeutics over the past decades have led to increasing survival rates for both paediatric and adult malignancies. Given the gonadotoxic effect of many cancer treatments, more women develop POF. Markers that predict whether women are at risk of POF would, therefore, aid in early diagnosis and fertility counselling.

The history of past and present status has been taken in our research. Women on the process of natural aging and disease-induced ovarian aging are all included. The key factors that influence ovary aging may be identified by epidemiological and molecular biological research.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Statue ≥ 70,
* WBC > 3,000/mm³,
* Hb > 9.0g/dl,
* Platelet > 100,000 /mm³,
* SGOT/SGPT < 60 IU/L,
* T-Bil < 1.5 mg/dL,
* Cr < 1.2 mg/dL,
* PaO2 > 80 torr,
* normal ECG,
* Written informed consent.

Exclusion Criteria:

* Patients without information,
* clinical risk factors,
* Patients who have active infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with normal ovarian function or decreased ovarian function
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
ovarian function evaluation including parameters FSH(mIu/ml), LH(mIu/ml), E2(pg/ml), T(ng/dl) for individuals with normal ovarian function (more than 2 000 women) and ovarian failure(more than 1 000 women). | up to 3 year
  FSH(mIu/ml), LH(mIu/ml), E2(pg/ml), T(ng/dl) levels were measured using a chemiluminescence-based immunometric assay on an ADVIA Centaur immunoassay system (Siemens Healthcare Diagnostics Inc., Tarrytown, NY, USA).

SECONDARY OUTCOMES:
women's reproductive function including pregnancy rate | up to 3 year
  pregnancy rate was recorded once a year

OTHER OUTCOMES:
ovarian function including parameters FSH(mIu/ml), LH(mIu/ml), E2(pg/ml) and T(ng/dl) and reproductive function including pregnancy rate after treatment for young female patients who have benign or malignant tumor | up to 3 year
  FSH(mIu/ml), LH(mIu/ml), E2(pg/ml) and T(ng/dl) levels were measured using a chemiluminescence-based immunometric assay on an ADVIA Centaur immunoassay system (Siemens Healthcare Diagnostics Inc., Tarrytown, NY, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, MD.PHD., Study Chair — Huazhong University of Science and Technology
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Wen J, Huang K, Du X, Zhang H, Ding T, Zhang C, Ma W, Zhong Y, Qu W, Liu Y, Li Z, Deng S, Luo A, Jin Y, Zhang J, Wang S. Can Inhibin B Reflect Ovarian Reserve of Healthy Reproductive Age Women Effectively? Front Endocrinol (Lausanne). 2021 Apr 14;12:626534. doi: 10.3389/fendo.2021.626534. eCollection 2021. PMID 33935966
- [Derived] Du X, Ding T, Zhang H, Zhang C, Ma W, Zhong Y, Qu W, Zheng J, Liu Y, Li Z, Huang K, Deng S, Ma L, Yang J, Jiang J, Yang S, Huang J, Wu M, Fang L, Lu Y, Luo A, Wang S. Age-Specific Normal Reference Range for Serum Anti-Mullerian Hormone in Healthy Chinese Han Women: A nationwide Population-Based Study. Reprod Sci. 2016 Aug;23(8):1019-27. doi: 10.1177/1933719115625843. Epub 2016 Jan 13. PMID 26763552